CLINICAL TRIAL: NCT04495660
Title: Restauration of the Auditory and Cognitive Functions in Cochlear Implanted Deaf Children in FNIRS
Acronym: HearCog
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC31/18/0047
Record Dates: First submitted 2020-06-04; First posted 2020-08-03 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Deafness
Keywords: Functional Neuroimaging; Profound and Severe Hearing Loss; Cochlear implant
MeSH Terms: conditions — Deafness; Hearing Loss | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Severe/profoundly deaf children 10-24 months old (Experimental): The cohort 1 includes patients aged 10-24 months old about to be implanted
  Interventions: Device: Near InfraRed Spectroscopy (fNIRS); Behavioral: Passive perceptual stimulation; Behavioral: Task A not B; Behavioral: VSWMT task; Behavioral: The sensory room
- Severe/profoundly deaf children 3-7 years old (Experimental): The cohort 2 includes 3-7 years old cochlear implanted patients (implanted before 24 months of age)
  Interventions: Device: Near InfraRed Spectroscopy (fNIRS); Behavioral: Passive perceptual stimulation; Behavioral: VSWMT task; Behavioral: Perceptual Go-No-Go; Behavioral: Verbal memory task
- Normally hearing children 10-24 months old (Other): The cohort 1 includes patients aged 10-24 months matched in age and sex with normally hearing children
  Interventions: Device: Near InfraRed Spectroscopy (fNIRS); Behavioral: Passive perceptual stimulation; Behavioral: Task A not B; Behavioral: VSWMT task; Behavioral: The sensory room
- Normally hearing children 3-7 years old (Other): The cohort 2 includes 3-7 years old matched in sex and age with cochlear implanted patients
  Interventions: Device: Near InfraRed Spectroscopy (fNIRS); Behavioral: Passive perceptual stimulation; Behavioral: VSWMT task; Behavioral: Perceptual Go-No-Go; Behavioral: Verbal memory task

INTERVENTIONS:
Device: Near InfraRed Spectroscopy (fNIRS) — Functional neuroimaging examination by fNIRS at each follow-up visit for all children of both cohorts: this non-invasive imaging technique involves the installation of a cap carrying electrodes to collect brain activity on the surface of the scalp , during stimulation. It is very insensitive to movement and therefore represents a method particularly suitable for its use in children. In addition, this technique is compatible with the cochlear implant. It will be used during 6 tasks adapted to each cohort
Behavioral: Passive perceptual stimulation — Passive perceptual stimulation: For this passive task the child is on his parents' lap in front of a screen. He will see images, hear everyday noises and watch small videos. Duration 8-10 minutes.
Behavioral: Task A not B — Task A not B: the child will play with an adult who will hide an object under a cloth several times. The child will have to find the hidden object. Duration 10 minutes maximum
  Arms: Normally hearing children 10-24 months old; Severe/profoundly deaf children 10-24 months old
Behavioral: VSWMT task — VSWMT task: the child will be on the parents' lap in front of a screen and will watch a monkey hiding bananas in the trees several times. Duration of 10 minutes maximum.
Behavioral: Perceptual Go-No-Go — Perceptual Go-No-Go: This perceptual task consists in the discrimination of images (faces) and sounds (words) through 3 conditions (auditory, visual and visuo-auditory) presented independently of each other and lasts 15 to 20 minutes in total. It is presented by means of a computer
  Arms: Normally hearing children 3-7 years old; Severe/profoundly deaf children 3-7 years old
Behavioral: Verbal memory task — Verbal memory task :the child will be presented with 5 lists of 5 words which he will have to restore after a predefined delay of a few seconds. Its duration does not exceed 10 minutes.
  Arms: Normally hearing children 3-7 years old; Severe/profoundly deaf children 3-7 years old
Behavioral: The sensory room — The sensory room: the child will sit in the middle of a carpet and play with the adult. He will hear everyday noises and see light effects. Duration 8-10 minutes
  Arms: Normally hearing children 10-24 months old; Severe/profoundly deaf children 10-24 months old

SUMMARY:
The principal aim of this study is to evaluate the cortical developement of perceptual skills and executive functions over time, in children with cochlear implants aged 10-24 months and 3-7 years compared with normally hearing subjects (NHS). To do this, the investigator will use functional Near InfraRed Spectroscopy (fNIRS) during 4 tasks that engage the childs perceptual and cognitive skills over a period of 18 months. The performance scores obtained by each participants as well as the cortical activity will be analysed and decrypted.

DETAILED DESCRIPTION:
When confronted with a severe to profound congenital bilateral hearing loss, cochlear implantation is considered to be the preferential treatment method as it restaures auditory function and enables language acquisition for communication purposes. When cochlear implantation is done before 2 and a half years old, better results are obtained in terms of language, communication and social developement, as well as reading skills. However when a cochlear implantation occurs between 2 and 5 years of age, speech and language skills do develop but communication and reading skills are altered. Therefore, when a cochlear implant is placed before the age of 2 and a half we find ourselves within the maximal cerebral plasticity window for speech, language and communication developement.

This study is divided into two cohorts, the first aged 10-24 months and the second 3-7 years. All children will be seen for 5 sessions, spread out at regular intervals, over a period of 18 months and will participate in two perceptual tasks and two cognitive tasks. The children will also have a speech and language assessment at T-0 and T+12. The cochlear implanted patients will continue to be seen by the ENT service and the sessions will be organised to coincide with their natural follow up. As it is a non-interventional study, no follow-up would be needed. After the study patients will continue to receive the same quality of care.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

Cohort 1 :

* 10-24 months old children will be included.
* All participants have to be affiliated to the social health security system and parental consent is obligatory.
* All congenitally deaf patients will have a severe to profound hearing loss and about to be fitted with a cochlear implant.
* Normally hearing counterparts shall have normal hearing as evidenced by acoustical otoemissions (AOE) in both ears.

Cohort 2 :

* 3-7 years old children will be included.
* All participants have to be affiliated to the social health security system and parental consent is obligatory.
* All congenitally deaf patients will have a cochlear implant, and they will have been implanted before 2 years of age.
* Normally hearing counterparts shall have normal hearing as evidenced by acoustical otoemissions (AOE) in both ears.

Exclusion Criteria:

* Exclusion criteria include psycho-neurological diseases, other sensorineural or motor deficiency, familial bilingualism, medications affecting vigilance and child whose both parents benefit from a legal protection measure

Ages: 10 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2026-06-03 (Estimated)

PRIMARY OUTCOMES:
Evolution of Oxyhemoglobin (O2Hb) measure | 60 months
  Oxyhemoglobin (O2Hb) rates measured on the auditory cortex during an auditory stimulus.
Evolution of Deoxyhemoglobin (HHb) measure | 60 months
  Deoxyhemoglobin (HHb) rates measured on the auditory cortex during an auditory stimulus.

SECONDARY OUTCOMES:
Activation of the cortical area for children with normal hearing and children benefiting from CI | 60 months
  Describe the evolution of the perceptual capacities of children benefiting from CI, compared to the typical development in children with normal hearing
Look the executive function when performing tasks describe in Arms and intervention chapter, between children with normal hearing and children benefiting from CI | 60 months
  Describe the evolution of the executive functions of children benefiting from CI, compared to the typical development in normal hearing children
Correlation of link between the evolution of perceptual hearing skills and the development of post-implantation language skills. | 60 months
  Evolution of language.
Make activation cards of the cortical reorganization between these two groups | 60 months
  Describe the cortical reorganization of the auditory area post implantation. performances obtained during perceptual anc cognitive tasks
Make activation cards of the cortical reorganization between these two groups | 60 months
  Describe the cortical reorganization of the visual area post implantation. performances obtained during perceptual anc cognitive tasks
Comparison | 60 months
  Correlation of link between cortical activation in post-implantation fNIRS and:
  * perceptual and executive functions over time in deep deaf children after CI;
  * language skills over time in deep deaf children after CI.

CONTACTS AND LOCATIONS:
Overall Officials: Yohan GALLOIS, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Gallois Yohan, Toulouse, France

IPD SHARING:
Plan to Share IPD: No